CLINICAL TRIAL: NCT00123136
Title: Bi-Axial Rotating Magnetic Field Therapy in Refractory Neuropathic Foot Pain Secondary to Diabetic Peripheral Neuropathy. Multi-Center, Randomized Placebo Controlled Trial
Brief Title: Bi-Axial Rotating Magnetic Field Therapy in Refractory Neuropathic Foot Pain Secondary to Diabetic Peripheral Neuropathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Weintraub, Michael I., MD, FACP, FAAN (Individual)
Collaborators: Nu-Magnetics Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-81440-DPN
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2006-07-04 (Estimated); Status verified 2006-06

CONDITIONS: Diabetic Neuropathies
Keywords: pulsed magnetic field therapy; diabetic peripheral neuropathy; neuromodulation; diabetic peripheral neuropathic pain; sleep benefit; diabetic peripheral neuropathic functioning
MeSH Terms: conditions — Diabetic Neuropathies

INTERVENTIONS:
Device: foot energizer

SUMMARY:
The researchers will study the application of a commercial pulsed magnetic stimulating device to the feet of patients with moderate-severe foot pain secondary to diabetic peripheral neuropathy (DPN).

ELIGIBILITY:
Inclusion Criteria:

* DPN stage 2 and 3; symptomatic > 6 months

Exclusion Criteria:

* Pacemaker in patient or mate

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2005-08; Study Completion 2006-12

PRIMARY OUTCOMES:
reduction of neuropathic foot pain
improve quality of life

SECONDARY OUTCOMES:
serial changes in EDX, QST, autonomic functions, biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Michael Weintraub, MD, Principal Investigator — New York Medical College
Locations (1):
- Michael I. Weintraub MD 325 S. Highland Avenue, Briarcliff, New York, United States

REFERENCES:
- [Derived] Weintraub MI, Herrmann DN, Smith AG, Backonja MM, Cole SP. Pulsed electromagnetic fields to reduce diabetic neuropathic pain and stimulate neuronal repair: a randomized controlled trial. Arch Phys Med Rehabil. 2009 Jul;90(7):1102-9. doi: 10.1016/j.apmr.2009.01.019. PMID 19577022